CLINICAL TRIAL: NCT00297674
Title: Clarithromycin as Immunomodulatory Therapy for the Management of Septic Syndrome by Ventilator-Associated Pneumonia
Brief Title: Intravenous Clarithromycin in Septic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACA-GREC-2004-01
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2006-02-28 (Estimated); Status verified 2004-07

CONDITIONS: Sepsis; Ventilator Associated Pneumonia
Keywords: clarithromycin; sepsis; immunomodulation
MeSH Terms: conditions — Sepsis; Pneumonia, Ventilator-Associated

INTERVENTIONS:
Drug: Intravenous Clarithromycin

SUMMARY:
The aim of this clinical trial is to clarify the clinical efficacy of clarithromycin as immunotherapy for the management of septic syndrome by ventilator-associated pneumonia.

DETAILED DESCRIPTION:
The rationale of the trial is based on the favorable results of experimental studies of sepsis by multidrug-resistant Pseudomonas aeruginosa and by susceptible Escherichia coli in rabbits where clarithromycin was administered intravenously. Data from these latter studies suggest that administration of clarithromycin extended survival and attenuated systemic inflammatory response. Their major endpoint was successful immunotherapy achieved when clarithromycin was administered on presentation of symptoms of sepsis-induced pulmonary edema; on the contrary, former clinical trials for immunotherapies of sepsis were based on animal studies where the under evolution immunomodulator was administered before bacterial challenge. The efficacy of administration of clarithromycin upon presentation of septic syndrome in animal studies, renders its application promising in the clinical field.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent provided by first or second degree relatives;
2. intubation and mechanical ventilation at least 48 hours prior to enrolment; c) age of patients equal to or more than 18 years;

d) diagnosis of Ventilator Associated Pneumonia; and e) signs of sepsis

Exclusion Criteria:

1. neutropenia, defined as less than 500 neutrophils/mm3;
2. HIV infection;
3. oral intake of corticosteroids at a dose equal to or higher than 1mg/kg equivalent prednisone for a period greater than one month;
4. administration of drotrecogin alpha the last five days prior to enrolment; and e) atrioventricular block of second or third degree.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-06; Study Completion 2005-12

PRIMARY OUTCOMES:
Estimation of crude mortality by any reason of each study group
Estimation of attributable mortality by VAP of each study group
7-day mortality rate of each group
28-mortality rate of each group
Rate of progression to multiple organ failure and septic shock (and number of failing organs) of each study group
Time to progression to multiple organ failure and septic shock of each study group
Days of resolution of VAP
Days in ICU after diagnosis of VAP

SECONDARY OUTCOMES:
Influence of administration of clarithromycin on systemic inflammatory response

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J Giamarellos-Bourboulis, MD, PhD, Study Chair — University of Athens, Medical School, Greece; Helen Giamarellou, MD, PhD, Principal Investigator — University of Athens, Medical School, Greece; Apostolos Armaganidis, MD, PhD, Principal Investigator — University of Athens, Medical School, Greece; Charis Roussos, MD, PhD, Principal Investigator — University of Athens, Medical School, Greece
Locations (3):
- Greece (3):
  - 1st Department of Critical Care, Evangelismos General Hospital, Athens
  - 2nd Department of Critical Care, ATTIKON University Hospital, Athens
  - 4th Department of Internal Medicine, ATTIKON University Hospital, Athens

REFERENCES:
- [Background] Giamarellos-Bourboulis EJ, Adamis T, Laoutaris G, Sabracos L, Koussoulas V, Mouktaroudi M, Perrea D, Karayannacos PE, Giamarellou H. Immunomodulatory clarithromycin treatment of experimental sepsis and acute pyelonephritis caused by multidrug-resistant Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2004 Jan;48(1):93-9. doi: 10.1128/AAC.48.1.93-99.2004. PMID 14693524
- [Background] Giamarellos-Bourboulis EJ, Baziaka F, Antonopoulou A, Koutoukas P, Kousoulas V, Sabracos L, Panagou C, Perrea D, Giamarellou H. Clarithromycin co-administered with amikacin attenuates systemic inflammation in experimental sepsis with Escherichia coli. Int J Antimicrob Agents. 2005 Feb;25(2):168-72. doi: 10.1016/j.ijantimicag.2004.08.018. PMID 15664488
- [Background] Giamarellos-Bourboulis E, Adamis T, Sabracos L, Raftogiannis M, Baziaka F, Tsaganos T, Koutoukas P, Plachouras D, Karayannacos P, Giamarellou H. Clarithromycin: immunomodulatory therapy of experimental sepsis and acute pyelonephritis by Escherichia coli. Scand J Infect Dis. 2005;37(1):48-54. doi: 10.1080/00365540510026832. PMID 15764190
- [Derived] Vittoros V, Kyriazopoulou E, Lada M, Tsangaris I, Koutelidakis IM, Giamarellos-Bourboulis EJ. Soluble fms-like tyrosine kinase 1, placental growth factor and procalcitonin as biomarkers of gram-negative sepsis: Analysis through a derivation and a validation cohort. Medicine (Baltimore). 2021 Nov 5;100(44):e27662. doi: 10.1097/MD.0000000000027662. PMID 34871241
- [Derived] Karakike E, Kyriazopoulou E, Tsangaris I, Routsi C, Vincent JL, Giamarellos-Bourboulis EJ. The early change of SOFA score as a prognostic marker of 28-day sepsis mortality: analysis through a derivation and a validation cohort. Crit Care. 2019 Nov 29;23(1):387. doi: 10.1186/s13054-019-2665-5. PMID 31783881
- [Derived] Strouvalis I, Routsi C, Adamopoulou M, Raftogiannis M, Renieris G, Orfanos SE, Kotanidou A, Sabracos L, Giamarellos-Bourboulis EJ. Early increase of VEGF-A is associated with resolution of ventilator-associated pneumonia: Clinical and experimental evidence. Respirology. 2018 Oct;23(10):942-949. doi: 10.1111/resp.13320. Epub 2018 May 9. PMID 29741298
- [Derived] Tsaganos T, Raftogiannis M, Pratikaki M, Christodoulou S, Kotanidou A, Papadomichelakis E, Armaganidis A, Routsi C, Giamarellos-Bourboulis EJ. Clarithromycin Leads to Long-Term Survival and Cost Benefit in Ventilator-Associated Pneumonia and Sepsis. Antimicrob Agents Chemother. 2016 May 23;60(6):3640-6. doi: 10.1128/AAC.02974-15. Print 2016 Jun. PMID 27044546
- [Derived] Giamarellos-Bourboulis EJ. Immunomodulatory therapies for sepsis: unexpected effects with macrolides. Int J Antimicrob Agents. 2008 Nov;32 Suppl 1:S39-43. doi: 10.1016/j.ijantimicag.2008.06.004. Epub 2008 Aug 15. PMID 18707849